CLINICAL TRIAL: NCT05759117
Title: Prospective Evaluation of the Aetiologies, Management and Clinical Outcomes in Patients With Pleural Effusion
Brief Title: Prospective Evaluation of Patients With Pleural Effusion
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Clinical Lecturer, Chinese University of Hong Kong
Other Study IDs: ProspectivePleuralEffusion
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion | interventions — Thoracentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — 40mL pleural fluid will be collected during thoracentesis or pleural drain insertion, or from collecting bags. The research pleural fluid will be transferred on ice and stored at - 80oC until assay for subsequent approved studies.
  6mL blood will be collected. The blood will be centrifuged, and the supernatant will be stored at - 80oC until assay for subsequent approved studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pleural effusion: All patients with pleural effusion who will undergo thoracentesis
  Interventions: Procedure: thoracentesis

INTERVENTIONS:
Procedure: thoracentesis — A type of pleural procedure that will yield pleural fluid for subsequent analysis
  Other Names: chest drain insertion

SUMMARY:
Having a pleural effusion is a common reason for being hospitalized, as it usually requires in-patient care for invasive diagnostic and therapeutic procedures. Specific subtypes of pleural effusion may warrant recurrent admissions, a longer hospital stay and consume more healthcare resources. Despite the recent advancement of pleural medicine, better research is increasingly desired to fill the gaps in establishing an early diagnosis and optimal management of pleural effusion from various causes. Local data on different aspects of pleural effusion is also lacking.

DETAILED DESCRIPTION:
The aetiologies of pleural effusion range from cardio-respiratory diseases, malignancy, infection to systemic inflammatory conditions. However, data on the exact incidence of individual causes of pleural effusion is inadequate. Conflicting results on the aetiologies of pleural effusion were shown in several retrospective and prospective studies based in different geographical regions, which may be explained by the different epidemiology of common diseases in the corresponding areas and patients recruited. Despite a common clinical problem, the incidence and aetiology of pleural effusion have not been examined on a population level in Hong Kong. Therefore, a local study is necessary to inform physicians about the disease burden of pleural effusion.

The management of pleural disease can be heterogeneous, as reflected by a recent multi-institutional questionnaire study in Hong Kong. Infrequent updates of international guidelines of pleural medicine, lack of an established registry reflecting the patient burden, procedure load and complications may contribute. Delayed or suboptimal management of pleural diseases can lead to unnecessary invasive procedures, prolonged hospital stays and even higher mortality rates. A local registry should be established to stocktake and understand diagnostic accuracy and complication rates of pleural procedures and reflects the real-life practice by hospital physicians.

This prospective study aims at evaluating the aetiology and management of pleural diseases prospectively. The management by the attending doctors will not be interfered. Recruited patients will be divided into subgroups based on their characteristics for further analysis. The data collected from this study will guide the planning of subsequent research to overcome the knowledge and service gap in managing pleural diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for pleural effusion.
* Pleural tapping will be performed for pleural fluid analysis.
* Aged 18 years old or above

Exclusion Criteria:

- Failed to obtain informed consent due to the patient's refusal or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have pleural effusion and will undergo thoracentesis for pleural fluid sampling
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Aetiology of pleural effusion | 1 month
  spectrum of aetiology for pleural effusion

SECONDARY OUTCOMES:
Management of pleural effusion | 1 month
  common clinical practice of handling pleural effusion will be evaluated
Prognosis of pleural effusion | 1 month
  need for hospitalization, pleural procedure, complication rate and time required to establish a diagnosis for patients with pleural effusion will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Study Director — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Chinese University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No